CLINICAL TRIAL: NCT00326599
Title: A Randomized Phase II Study of Gemcitabine and Carboplatin With or Without AZD2171 as First-Line Therapy in Advanced Non-Small Cell Lung Cancer
Brief Title: Gemcitabine and Carboplatin With or Without AZD2171 as First-Line Therapy in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0528; NCI-2012-02694 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000468945 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; cediranib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, carboplatin IV over 30 minutes on day 1, and oral AZD2171 once daily on days 1-21. Treatment repeats every 21 days for up to 6 courses. Patients achieving stable disease, partial response, or complete response after 6 courses of therapy receive AZD2171 alone as above. Treatment with AZD2171 repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: cediranib maleate; Drug: gemcitabine hydrochloride
- Arm II (Active Comparator): Patients receive gemcitabine and carboplatin as in arm I. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: carboplatin — Given IV
Drug: cediranib maleate — Given orally
  Arms: Arm I
Drug: gemcitabine hydrochloride — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. AZD2171 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving gemcitabine and carboplatin together with AZD2171 may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well giving gemcitabine and carboplatin together with AZD2171 works compared to giving gemcitabine and carboplatin without AZD2171 as first-line therapy in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the objective tumor response rate in patients with stage IIIB or IV non-small cell lung cancer treated with gemcitabine hydrochloride, carboplatin, and AZD2171 as first-line therapy.

Secondary

* Compare the proportion of patients who are progression-free at 6 months after treatment with gemcitabine hydrochloride and carboplatin with vs without AZD2171.
* Compare the duration of response for responding patients treated with these regimens.
* Compare the time-to-progression and time-to-treatment failure.
* Compare the 1-year overall survival.
* Compare the clinical toxicities.
* Assess the safety and tolerability of these regimens in these patients.

Tertiary

* Collect blood and tumor specimens for future evaluation of pharmacogenetic and proteomic markers of tumor response and toxicity to therapy with these agents.
* Bank paraffin-embedded tissue blocks/slides and blood samples for future histochemistry evaluation and DNA extraction.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior adjuvant therapy (yes vs no) and ECOG performance status (0 vs 1). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, carboplatin IV over 30 minutes on day 1, and oral AZD2171 once daily on days 1-21. Treatment repeats every 21 days for up to 6 courses. Patients achieving stable disease, partial response, or complete response after 6 courses of therapy receive AZD2171 alone as above. Treatment with AZD2171 repeats every 21 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine and carboplatin as in arm I. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection periodically during study for pharmacologic correlative studies.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 102 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Squamous cell histology allowed
  * No mixed histology with small cell component
* Stage IIIB (with pleural effusion) or stage IV disease

  * Presence of peritoneal or pericardial effusion alone in the absence of cytologic evidence is not allowed
* Measurable disease, defined as ≥ 1 lesion with longest diameter ≥ 2.0 cm by conventional techniques OR ≥ 1.0 cm by spiral CT scan

  * If the only site of measurable disease was previously irradiated, progressive disease must be evident
* Ineligible for bevacizumab therapy
* No symptomatic, untreated, or uncontrolled CNS metastases

  * CNS metastases treated with whole-brain radiation (WBRT) allowed 4 weeks after completion of WBRT

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 3 times upper limit of normal (ULN)
* ALT and AST ≤ 3 times ULN (5 times ULN if liver involvement)
* Alkaline phosphatase ≤ 5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception
* No proteinuria ≥ 1+
* No uncontrolled blood pressure (BP), defined as systolic BP > 150 mm Hg and/or diastolic BP > 100 mm Hg in spite of adequate antihypertensive therapy
* No impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of AZD2171 (e.g., ulcerative disease, uncontrolled nausea, vomiting, or diarrhea, malabsorption syndrome, or small bowel resection)
* No seizure disorder
* No significant traumatic injury within 4 weeks prior to study entry
* No second primary malignancy except any of the following:

  * Carcinoma in situ of the cervix
  * Nonmelanoma skin cancer
  * Prior malignancy diagnosed and definitively treated ≥ 5 years ago with no subsequent evidence of recurrence
  * History of low-grade (Gleason score ≤ 6) localized prostate cancer even if diagnosed < 5 years prior to registration
  * Treated stage I breast cancer ≤ 5 years prior to registration
* No uncontrolled intercurrent illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Significant pulmonary symptoms at baseline due to disease
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements
  * Baseline hemoptysis
  * Cavitating lesions
* No QTc prolongation > 500 msec or other significant ECG abnormality within the past 14 days
* No New York Heart Association class III or IV disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for advanced lung cancer

  * Neoadjuvant or adjuvant therapy for lung cancer within the past 12 months allowed
* More than 12 months since prior immunotherapy and biologic therapy
* More than 4 weeks since prior radiotherapy (2 weeks for palliative radiotherapy to skeletal metastases)
* At least 2 weeks since prior WBRT
* No radiotherapy to ≥ 25% of bone marrow
* No major surgery (i.e., laparotomy) or open biopsy within 4 weeks prior to study entry (2 weeks for minor surgery)

  * Insertion of a vascular access device not considered major or minor surgery
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent grapefruit or grapefruit juice during AZD2171 treatment
* No concurrent drugs or biologics with proarrhythmic potential
* Concurrent palliative radiotherapy to nontarget sites (i.e., painful pre-existing bony metastasis) allowed with AZD2171 (chemotherapy is held until completion of radiotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex A. Adjei, MD, PhD, Study Chair — Roswell Park Cancer Institute
Locations (154):
- United States (154):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Mercy Hospital at Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Background] van Cruijsen H, Voest EE, van Herpen CM, et al.: Phase I evaluation of AZD2171, a highly potent, selective VEGFR signaling inhibitor, in combination with gefitinib, in patients with advanced tumors. [Abstract] J Clin Oncol 24 (Suppl 18): A-3017, 125s, 2006.
- [Result] Dy GK, Mandrekar SJ, Nelson GD, Meyers JP, Adjei AA, Ross HJ, Ansari RH, Lyss AP, Stella PJ, Schild SE, Molina JR, Adjei AA. A randomized phase II study of gemcitabine and carboplatin with or without cediranib as first-line therapy in advanced non-small-cell lung cancer: North Central Cancer Treatment Group Study N0528. J Thorac Oncol. 2013 Jan;8(1):79-88. doi: 10.1097/JTO.0b013e318274a85d. PMID 23232491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred-and one (101) participants were enrolled between June 15, 2007 and December 5, 2008. Data for this report were frozen on September 13, 2011.
Pre-assignment Details: Five participants were excluded from all analyses due to withdrew consent or never received study treatment: 1 lead-in arm I; 2 phase II arm I; and 2 phase II arm II. The starting cediranib dose of 45 mg was not tolerable and was reduced to 30 mg once daily on a continuous schedule for the phase II portion of the study.
Groups:
- Lead-in Phase: Arm I (Cediranib + Gemcitabine + Carboplatin): Patients receive oral cediranib 45mg once daily in combination with chemotherapy, gemcitabine 1000 mg/m2 on days 1 and 8 and carboplatin dosed to an area under the serum concentration time curve of 5 on day 1 via intravenous infusion every 3 weeks for a maximum of six cycles.
- Lead-in Phase: Arm II (Gemcitabine + Carboplatin); Phase II: Arm II (Gemcitabine + Carboplatin): Patients receive gemcitabine 1000 mg/m2 on days 1 and 8 and carboplatin dosed to an area under the serum concentration time curve of 5 on day 1 via intravenous infusion every 3 weeks for a maximum of six cycles.
- Phase II: Arm I (Cediranib + Gemcitabine + Carboplatin): Patients receive oral cediranib 30mg once daily in combination with chemotherapy, gemcitabine 1000 mg/m2 on days 1 and 8 and carboplatin dosed to an area under the serum concentration time curve of 5 on day 1 via intravenous infusion every 3 weeks for a maximum of six cycles.
Period: Overall Study
Arm/Group | Lead-in Phase: Arm I (Cediranib + Gemcitabine + Carboplatin) | Lead-in Phase: Arm II (Gemcitabine + Carboplatin) | Phase II: Arm I (Cediranib + Gemcitabine + Carboplatin) | Phase II: Arm II (Gemcitabine + Carboplatin)
Started | 6 | 3 | 58 | 29
Completed | 0 | 2 | 5 | 10
Not Completed | 6 | 1 | 53 | 19
Not completed — Withdrawal by Subject | 1 | 0 | 5 | 2
Not completed — Adverse Event | 1 | 0 | 32 | 3
Not completed — Disease Progression | 3 | 1 | 13 | 11
Not completed — Alternate Treatment | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 2
Not completed — Other Unspecified Reason | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lead-in Phase: Arm I (Cediranib + Gemcitabine + Carboplatin) | Lead-in Phase: Arm II (Gemcitabine + Carboplatin) | Phase II: Arm I (Cediranib + Gemcitabine + Carboplatin) | Phase II: Arm II (Gemcitabine + Carboplatin) | Total
Number analyzed (Participants) | 6 | 3 | 58 | 29 | 96
Age, Continuous [Median (Full Range); unit: years] | 65.5 [62 to 75] | 74 [64 to 76] | 65 [46 to 81] | 64 [45 to 82] | 64 [45 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 26 | 12 | 45
  Male | 2 | 0 | 32 | 17 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 2 | 5
  White | 6 | 3 | 55 | 26 | 90
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 58 | 29 | 96
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0=Asymptomatic and fully active | 3 | 1 | 33 | 17 | 54
  1=Symptomatic and fully ambulatory | 3 | 2 | 25 | 12 | 42
Before adjuvant treatment [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 2 | 1 | 4
  No | 5 | 3 | 56 | 28 | 92
Cell type [Count of Participants; unit: Participants]
  Squamous | 0 | 1 | 9 | 8 | 18
  Adenocarcinoma | 4 | 1 | 22 | 16 | 43
  All other | 2 | 1 | 27 | 5 | 35

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response Rate (Complete Response and Partial Response) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) (Phase II Patients Only)
Description: A confirmed tumor response was defined as a complete response (CR) or partial response (PR) noted as the objective status on 2 consecutive evaluations at least 6 weeks apart.
  Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria:
  * Complete Response (CR): disappearance of all target lesions;
  * Partial Response (PR) 30% decrease in sum of longest diameter of target lesions
Time Frame: Up to 5 years
Population: All phase II participants who met eligibility criteria and have received at least one cycle of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Arm I (Cediranib + Gemcitabine + Carboplatin) | Phase II: Arm II (Gemcitabine + Carboplatin)
Number analyzed (Participants) | 58 | 29
percentage of participants | 19 [10 to 31] | 20 [8 to 40]

2. Secondary Outcome: Progression-free Survival Rate at 6 Months After Randomization (Phase II Patients Only)
Description: Estimated using the Binomial point estimator (number of successes divided by the total number of evaluable patients). A patient is classified as a success if alive and progression-free at 6 months.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 6 months
Population: All phase II participants who met eligibility criteria and have received at least one cycle of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Arm I (Cediranib + Gemcitabine + Carboplatin) | Phase II: Arm II (Gemcitabine + Carboplatin)
Number analyzed (Participants) | 58 | 29
percentage of participants | 48 [35 to 62] | 38 [21 to 58]

3. Secondary Outcome: Progression-free Survival (Phase II Patients Only)
Description: Progression-free survival was defined as the time from study enrollment to the first date of disease progression or death as a result of any cause, whichever occurs first. Progression-free survival will be censored at the date of the last contact for patients who are still alive and who have not had disease progression.
Time Frame: Up to 5 years
Population: All phase II participants who met eligibility criteria and have received at least one cycle of treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Arm I (Cediranib + Gemcitabine + Carboplatin) | Phase II: Arm II (Gemcitabine + Carboplatin)
Number analyzed (Participants) | 58 | 29
months | 6.3 [4.7 to 7.9] | 4.5 [2.6 to 7.2]

4. Secondary Outcome: Time to Treatment Failure (Phase II Patients Only)
Description: Time to treatment failure was defined to be the time from date of registration to the date at which the patient was removed from the treatment due to progression, toxicity, refusal or death from any cause.
Time Frame: Up to 15 months
Population: All phase II participants who met the eligibility criteria and have ended the study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Arm I (Cediranib + Gemcitabine + Carboplatin) | Phase II: Arm II (Gemcitabine + Carboplatin)
Number analyzed (Participants) | 58 | 29
months | 2.48 [1.94 to 3.25] | 2.89 [1.71 to NA] — The upper limit of 95%CI was not attainable.

5. Secondary Outcome: Overall Survival at 1 Year After Randomization (Phase II Patients Only)
Description: Overall survival was defined as the time from study enrollment to the time of death from any cause. A patient is classified as a success if alive at 1 year.
Time Frame: 1 year
Population: All phase II participants who met eligibility criteria and started the treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Arm I (Cediranib + Gemcitabine + Carboplatin) | Phase II: Arm II (Gemcitabine + Carboplatin)
Number analyzed (Participants) | 58 | 29
percentage of participants | 48 [34.9 to 60.7] | 41 [23.7 to 58.3]

6. Secondary Outcome: Overall Survival (Phase II Patients Only)
Description: Overall survival was defined as the time from study enrollment to the time of death from any cause. Overall survival will be censored at the date of the last follow-up visit for patients who are still alive or lost to follow-up.
Time Frame: Up to 5 years
Population: All phase II participants who met eligibility criteria and started the treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Arm I (Cediranib + Gemcitabine + Carboplatin) | Phase II: Arm II (Gemcitabine + Carboplatin)
Number analyzed (Participants) | 58 | 29
months | 12.0 [7.5 to 20.6] | 9.9 [5.4 to 13.7]

7. Secondary Outcome: Dose Limiting Toxicity (DLT) (Lead-in Phase Arm I Patients Only)
Description: DLT was defined as an adverse event occurring in cycle 1 only, at least possibly attributed to the study treatment and meeting the following criteria: 1) Grade 4 absolute neutrophil count (ANC) >5 days or of any duration with fever >38.5 degree Celsius; 2) Grade 4 platelet count; 3) Grade 3 or higher non-hematologic toxicities (for nausea, vomiting or diarrhea, grade 3 toxicities will be DLT if they occur despite maximal use of anti-emetic support or anti-diarrhea agents, respectively); 4) Cediranib dose interruption of >14 days for drug-related toxicities.
Time Frame: Cycle 1 (up to 3 weeks)
Population: The first 6 participants treated on Arm I (lead-in phase).
Measure: Number; unit: participants
Arm/Group | Lead-in Phase: Arm I (Cediranib + Gemcitabine + Carboplatin)
Number analyzed (Participants) | 6
participants | 1

ADVERSE EVENTS:
Time Frame: Up to 15 months
Description: All participants who met eligibility criteria and started the treatment.
Arm/Group | Lead-in Phase: Arm I (Cediranib + Gemcitabine + Carboplatin) | Lead-in Phase: Arm II (Gemcitabine + Carboplatin) | Phase II: Arm I (Cediranib + Gemcitabine + Carboplatin) | Phase II: Arm II (Gemcitabine + Carboplatin)
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/3 | 39/58 | 8/29
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 58/58 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in Phase: Arm I (Cediranib + Gemcitabine + Carboplatin) (N=6) | Lead-in Phase: Arm II (Gemcitabine + Carboplatin) (N=3) | Phase II: Arm I (Cediranib + Gemcitabine + Carboplatin) (N=58) | Phase II: Arm II (Gemcitabine + Carboplatin) (N=29)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (5) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (1) | 11 (12) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 16 (20) | 4 (4)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 23 (28) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 7 (8) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in Phase: Arm I (Cediranib + Gemcitabine + Carboplatin) (N=6) | Lead-in Phase: Arm II (Gemcitabine + Carboplatin) (N=3) | Phase II: Arm I (Cediranib + Gemcitabine + Carboplatin) (N=58) | Phase II: Arm II (Gemcitabine + Carboplatin) (N=29)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (30) | 3 (16) | 53 (182) | 27 (95)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 11 (15) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (4) | 5 (8) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (6) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 4 (12) | 1 (2) | 32 (94) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2) | 1 (2) | 15 (22) | 2 (3)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (4) | 1 (1) | 16 (31) | 3 (4)
Nausea (Gastrointestinal disorders) | 2 (6) | 2 (7) | 35 (83) | 15 (30)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 1 (2) | 14 (22) | 6 (6)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 6 (28) | 3 (13) | 55 (202) | 26 (86)
Fever (General disorders) | 1 (1) | 0 (0) | 6 (6) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Leukocyte count decreased (Investigations) | 6 (27) | 3 (11) | 50 (129) | 23 (71)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Neutrophil count decreased (Investigations) | 6 (21) | 3 (7) | 45 (110) | 19 (54)
Platelet count decreased (Investigations) | 6 (19) | 3 (11) | 43 (101) | 23 (54)
Weight loss (Investigations) | 0 (0) | 0 (0) | 2 (8) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 8 (11) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (5) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (5) | 1 (5) | 13 (42) | 11 (23)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Taste alteration (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 15 (29) | 3 (4)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 2 (9) | 36 (99) | 19 (46)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (2) | 11 (18) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 3 (4) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 7 (18) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 12 (24) | 2 (3)
Hypertension (Vascular disorders) | 4 (16) | 3 (4) | 30 (67) | 4 (4)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 3 (4) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less